CLINICAL TRIAL: NCT05634161
Title: Usability of Cognitive Improvement Software in Cognitively Impaired Patients: Pilot Study
Status: Active, not recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, Jun Young Lee, Professor, Seoul National University Boramae Hospital
Other Study IDs: 20-2022-48
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cognitive Improvement software: Usability assessment of cognitive improvement software
  Interventions: Other: Cognitive improvement software

INTERVENTIONS:
Other: Cognitive improvement software — Cognitive improvement software

SUMMARY:
Usability study of software application that provide digitized cognitive intervention therapy for cognitively impaired patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients, 55~85 years
* Adequate vision, hearing and speaking for neuropsychological testing
* No difficulty in using mobile application using smartphone
* Patients with subjective memory complaints, confirmed by informants
* Cognitive impairment of SD 1 or greater from the age-adjusted normal range in Memory domain in CERAD-NP battery
* Global CDR 0.5 ~ 1
* Korean speaker
* Have an identified trial partner
* All subjects signed written consent

Exclusion Criteria:

* Those unable to provide consent
* History of transient ischemic attack, stroke, brain tumor
* History of diagnosis of major depression
* Symptoms that may interfere with the subject's testing procedure
* Cerebral hemorrhage
* Central nervous system infections
* Prohibited concomitant medication
* Known or suspected history of drug or alcohol abuse

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cognitively Impaired patients aged 55 to 85, based in South Korea.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Usability: Based on scenarios | Single-point evaluation (baseline)

SECONDARY OUTCOMES:
Usability: Based on user survey | Single-point evaluation (baseline)
Usability: Based on hemodynamic responses | Single-point evaluation (baseline)
Changes in Adas-cog | After 12 weeks of system usage
Changes in ADCS-ADL | After 12 weeks of system usage
Changes in self-reported quality of life | After 12 weeks of system usage
Changes in blood biomarker | After 12 weeks of system usage

OTHER OUTCOMES:
MMSE | Single-point evaluation (baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Young Lee, M.D., Ph.D., Principal Investigator — Department of Psychiatry, Seoul National University College of Medicine, Department of Psychiatry, SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea